CLINICAL TRIAL: NCT05783700
Title: Identification of Biomarkers for the Study of Sarcopenia and Its Evolution in Diabetic Patients.
Brief Title: Identification of Biomarkers for the Study of the Diabetic Foot and Evolution.
Acronym: SCFOOT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Esther Soler (Other)
Responsible Party: Sponsor-Investigator, Esther Soler, Bachelor of Science in Nursing, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: PI 138/2022
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus; Diabetic Foot; Sarcopenia; Neuropathy, Diabetic; Vascular Disease, Peripheral; Metabolic Syndrome
Keywords: DIABETES MELLITUS; DIABETIC FOOT; SARCOPENIA; NEUROPATHY, DIABETIC; VASCULAR DISEASE, PERIPHERAL
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Sarcopenia; Diabetic Neuropathies; Peripheral Vascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DIABETIC: PERFORMANCE OF BIOIMPEDANCIOMETRY WITH DETERMINATION OF:
  * Daily calorie intake
  * Body fat mass and percentage
  * Segmental body fat percentage
  * Resting Heart Rate
  * Lean Mass
  * Risk of sarcopenia
  * Proteins
  * Extra Cellular Water
  * Intracellular Water
  * Phase Angle
  * Visceral fat
  * Muscle mass
  * Segmental muscle mass
  * Muscle quality score
  * Total body water (%)
  * Metabolic age
  Interventions: Diagnostic Test: BIOIMPEDANCEMETRY

INTERVENTIONS:
Diagnostic Test: BIOIMPEDANCEMETRY — The impedance of cellular tissue can be modeled as a resistor (representing the extracellular path) in parallel with a resistor and capacitor in series (representing the intracellular path, the resistance that of intracellular fluid and the capacitor the cell membrane). This results in a change in impedance versus the frequency used in the measurement. Whole body impedance measurement is generally measured from the wrist to the ipsilateral ankle and uses either two (rarely) or four (overwhelmingly) electrodes. In the 2-elctrode (bipolar) configuration a small current on the order of 1-10 μA is passed between two electrodes, and the voltage is measured between the same whereas in the tetrapolar arrangement resistance is measured between as separate pair of proximally located electrodes. The tetrapolar arrangement is preferred since measurement is not confounded by the impedance of the skin-electrode interface

SUMMARY:
The European Working Group on Sarcopenia in the Elderly1 defines sarcopenia as a disorder of the progressive and generalized musculoskeletal system [1], which is associated with the increase and probability of adverse outcomes including falls, fractures, physical disability, and mortality [2]. what is associated with increased and likelihood of adverse outcomes including falls, fractures, disability physical and mortality [2]. For a long time, sarcopenia was associated with aging, affecting onlyold people. At present and after several research works related to fragility and theaging, it has been identified that the development of sarcopenia begins earlier in life [3], and that there are many contributing causes besides aging [4], [5]. This new knowledge has implications in the intervention of sarcopenia that prevents or delays its development. Sarcopenia is currently considered a muscle disease (muscle failure), based on adverse changes in the muscles of the musculoskeletal system accumulated throughout life, with loss of muscle strength such as main determinant [6], [7]. Sarcopenia has been overlooked in clinical practice, apparently due to to the complexity in determining the variables to be measured, how to measure them, and the values or cut-off points can guide diagnosis and treatment, and how best to assess the effects of therapeutic intervention [8]. In terms economic, the presence of sarcopenia increases the risk of hospitalization and increases the cost of care during hospital admission [9]. Diabetes is the main cause of non-traumatic amputation of the lower limb (MI), being foot ulcers diabetic the cause of 80% of the amputations of people with diabetes[10]. A study conducted by the Chongqing University Hospital showed that sarcopenia is independently related to the foot diabetic and that patients with diabetic foot have a worse prognosis if they suffer from sarcopenia. HYPOTHESIS: The surface electromyography (EMGs) signal recording of the foot musculature, will allow extracting biomarkers that allow monitoring and follow-up of sarcopenia in diabetic patients.

MAIN OBJECTIVES: 1- Generate tools based on artificial intelligence (AI) using the database with the biomarkers obtained, in order to analyze the predisposing and triggering risk factors associated with diabetic foot ulcers, according to the IWGDF2. 2- Describe the profile of the diabetic patient in terms of degree of sarcopenia with respect to the population without diabetes in a group of adults. DESIGN: Observational study comparison between cases and controls: a group with the presence of Diabetes Mellitus and another without. SAMPLE: Approximately 16% of diabetic patients will develop an ulcer during their evolution and the Annual incidence is 2-3%, which doubles to 6% in the presence of polyneuropathy. Population of the Department of Health 168,978. Prevalence of diabetes in Spain 7.8%. It is estimated that there are 13,182 in the department people with diabetes. Confidence level 95%, expected frequency of ulcers 6% and confidence limit 9%, it was calculates the sample of 26 patients. 30 patients per group will be recruited. GROUP 1: 30 patients with Diabetes Mellitus. GROUP 2: 30 control patients without Diabetes Mellitus. The period of inclusion of patients is estimated at 5 months. METHOD: the assessment interventions will be carried out in two days. During the first visit, examination to identify risk to the foot: clinical history (PA, comorbidity data, previous injuries to the feet).

feet..), examination of the vascular state, examination of loss of protective sensitivity, perception of pressure, skin inspection, inspection of bone/joint structures, physical limitations and level of knowledge of the foot care. During the second visit: diagnostic tests for sarcopenia (bioimpedance and electromyography), arthropometric measurements, malnutrition, dependence and activity marker tests.

EXPECTED RESULTS: clarify some aspects related to the sarcopenia-diabetic foot binomial, and isolate risk factors for future prevention, by obtaining biomarkers with EMGs in lower limbs.

DETAILED DESCRIPTION:
The European Working Group on Sarcopenia in the Elderly3 defines sarcopenia as a disorder of the progressive and generalized musculoskeletal system [1], which is associated with the increase and probability of adverse outcomes including falls, fractures, physical disability, and mortality [2]. During For a long time, sarcopenia was associated with aging, affecting only older people. currently and After various research papers related to frailty and aging, it has been identified that the development of sarcopenia begins earlier in life [3], and that there are many contributing causes to it in addition to aging [4], [5]. This new knowledge has implications for the intervention of the sarcopenia that prevents or delays its development. Sarcopenia is currently considered a muscle disease (muscle failure), based on adverse changes in the muscles of the muscular system skeletal muscle accumulated throughout life, with loss of muscle strength as the main determinant [6], [7].

Sarcopenia has been overlooked in clinical practice, apparently due to the complexity in determining the variables to be measured, how to measure them, and the values or cut-off points can guide a diagnosis and its treatment, and how best to assess the effects of therapeutic intervention [8]. In economic terms, the presence of sarcopenia increases the risk of hospitalization and increases the cost of care during admission hospital [9]. Diabetes is the main cause of non-traumatic amputation of the lower limb (MI), being foot ulcers diabetic the cause of 80% of the amputations of people with diabetes[10]. A study conducted by the Chongqing University Hospital showed that sarcopenia is independently related to the foot diabetic and that patients with diabetic foot have a worse prognosis if they suffer from sarcopenia. The percentage of patients with sarcopenia in diabetic foot is more than double that in patients without diabetic foot disease (EPD) (35.3% vs. 16.4%, P<0.001)[11]. The 5-year mortality rate in amputations of the MMI it is almost double in patients with sarcopenia than without sarcopenia (60.7% vs. 36.4%, P<0.006). There are three causes of PDE, peripheral arterial disease (PAD), diabetic neuropathy, and infection, and here the importance that sarcopenia has in this problem appears, because it accelerates its evolution. Yes ok the reasons are not well known about this link, there is something that is known, and that is that both neuropathy as vascular disease are associated with sarcopenia. Drey et al showed in a cross-sectional study, older adults with sarcopenia are more likely to lose motor neurons than those without sarcopenia loss of muscle mass [12]. Prior and her team provided evidence that sarcopenia in the elderly is associated with less capillarization. The authors also found that patients with sarcopenia presented higher proportion of neuropathy and EPD. It is for all of the above that neuropathy and vascular lesions could associate sarcopenia with diabetic foot [13]. The molecular bases of EPD-associated sarcopenia have not been clearly identified. However, it is known that the myokines and myometabolites that are normally released by muscle to connect with other organs and promote health, are altered. there is even knowledge evidence that a sarcopenic muscle has an overproduction of free radicals of oxygen (ROS) and nitrogen, something that is claimed to mediate neuropathy and vascular lesions, all of which could show the link between sarcopenia and EPD. So then, if it is indeed ensured that the loss of muscle mass is related to EPD, treating sarcopenia and its prevention, could be important for the prevention of the lesions

ELIGIBILITY:
Inclusion Criteria:

1. The sample will include all the people who sign the informed consent.
2. Patients aged between 18 and 80 years.
3. Patients diagnosed with Type 2 Diabetes Mellitus (more than 5 years from diagnosis), who continue to be monitored in the diabetes nursing office of the Health Department of the General Hospital of Elche.
4. Patients with Risk Level 0, Risk 1 and 2 according to the International Working Group on the Diabetic Foot -IWGDF.
5. Patient with control analysis, a maximum of one month prior to inclusion.

Exclusion Criteria:

1. People who do not give their consent to participate in the study.
2. Participants excluded for having problems walking (they used a cane or walker and/or had disabilities to stand up on their own)
3. Patients who have previously had treatment with plantar orthoses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients assisted at the San Fermín Specialty Center of the Elche General Hospital Health Department, with and without Type 2 Diabetes Mellitus.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2023-12-04 (Estimated); Study Completion 2024-01-07 (Estimated)

PRIMARY OUTCOMES:
BIOIMPEDANCEMETRY | FIFTEEN MINUTES
  Bioelectrical impedance analysis (BIA) is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Most body water is stored in muscle. Therefore, if a person is more muscular there is a high chance that the person will also have more body water, which leads to lower impedance. Since the advent of the first commercially available devices in the mid-1980s the method has become popular owing to its ease of use and portability of the equipment. It is familiar in the consumer market as a simple instrument for estimating body fat. BIA[1] actually determines the electrical impedance, or opposition to the flow of an electric current through body tissues which can then be used to estimate total body water (TBW), which can be used to estimate fat-free body mass and, by difference with body weight, body fat.

SECONDARY OUTCOMES:
Body fat mass and percentage | ONLY ONCE. 10 MINUTES
  Body fat mass is the weight of fat on your body. Body fat percentage is the weight of body fat mass in relation to total body weight.
  Body fat performs important functions, such as keeping the body warm or protecting the organs. It's important, but too much or too little fat is counterproductive to your health. A high percentage of fat can lead to lifestyle-related diseases such as type 2 diabetes or obesity, while a low percentage of fat can lead to osteoporosis, irregular menstruation, or loss of bone mass. Body analysis helps measure body fat percentage by calculating your body fat in relation to your total body weight. Too low a percentage means that the patient probably needs to make changes to their diet and exercise regimen to increase their fat mass to a healthier level, while a high percentage means they could benefit from more exercise and a healthier diet.
Segmental body fat percentage | ONLY ONCE. 10 MINUTES
  Measurement of body fat percentage by body part. By measuring the variation in fat percentages in both arms, both legs, and the torso separately, you can specifically monitor the effectiveness of your efforts and make adjustments as needed.
Visceral fat | ONLY ONCE. 10 MINUTES
  Visceral fat is found deep in the center of the abdomen. This fat surrounds and protects vital organs, such as the liver, pancreas, and kidneys.
  Visceral fat is found inside the muscular wall in the trunk of the body and protects vital organs. Visceral fat is not visible on the outside of the body and cannot be expressed. In addition to a healthy overall body fat percentage, it's important to keep a close eye on the amount of visceral fat. Especially as you get older. Too much visceral fat can lead to serious health problems, such as cardiovascular disease, type 2 diabetes, or high blood pressure.
Muscle mass | ONLY ONCE. 10 MINUTES
  Muscle mass includes skeletal muscle, smooth muscle (such as heart and digestive muscles) and the water in your muscles. Muscles act as the engine for your energy expenditure. As your muscle mass increases, the rate at which you burn energy (calories) increases. This speeds up your basal metabolic rate (BMR) and helps to reduce excess body fat. This is how you lose weight in a healthy way.
  A high muscle mass can reduce the risk of developing diabetes in adulthood. More skeletal muscle mass means more insulin receptor sites, which help with the uptake and regulation of glucose (sugar) deposited in the bloodstream after eating. 80% of glucose uptake takes place in skeletal muscle.
Muscle quality score | ONLY ONCE. 10 MINUTES
  Some people have huge muscles but can't lift much. It's not just quantity that counts when it comes to your muscles, quality matters a lot too. Even within your own body, the quality of your muscles can differ. If, for example, your left arm has better quality muscles than your right, an imbalance in your body is lurking. This in turn can lead to injury. From the age of 18 it is possible to evaluate the quality of your muscles. This is assessed on the basis of the relationship between muscle mass and height.
Total body water (%) | ONLY ONCE. 10 MINUTES
  Body water percentage is the amount of fluid in the body, expressed as a percentage of total body weight.
  Water plays an important role in various bodily processes and is found in every cell, tissue and organ. A healthy body water percentage for women is between 45% and 60%. For men, it is between 50% and 65%.
  A healthy percentage of body fluids reduces the risk of health problems and ensures that the body functions properly.
  The body's water content is constantly changing. Water is lost through urine, sweat and breathing, but your hydration level can also vary depending on, for example, alcohol consumption, the flu or menstruation.
  The percentage of total body fluids decreases as the percentage of body fat increases. A person with a high body fat percentage may fall below the average body water percentage.
Bone mass | ONLY ONCE. 10 MINUTES
  Sarcopenia is currently considered a muscle disease (muscular failure), based on adverse changes in the muscles of the musculoskeletal system accumulated throughout life, with loss of muscle strength as the main determinant. A study conducted by Chongqing University Hospital showed that sarcopenia is independently related to diabetic foot and that patients with diabetic foot have a worse prognosis if they have sarcopenia.
  Sarcopenia is more frequent in patients with Type 2 Diabetes Mellitus (DM2), without fully clarifying the direction of this association. Both share several pathogenic mechanisms, the most relevant being the insulin resistance characteristic of DM2, which could also alter the effect of insulin on muscle cell protein synthesis.
ONLY ONCE. 10 MINUTES | ONLY ONCE. 10 MINUTES
  BMR (Basal Metabolic Rate) is the minimum amount of energy or calories your body requires daily to function effectively when you are at rest. This includes sleep.
  Basal metabolic rate (BMR) is the minimum daily level of energy or calories your body requires at rest for your respiratory and circulatory organs, neural system, liver, kidneys, and other organs to function. effectively. Your BMR is heavily influenced by how much muscle you have. Increasing muscle mass increases your BMR, which increases the number of calories consumed and subsequently decreases the amount of body fat.
Body Mass Index | ONLY ONCE. 10 MINUTES
  A standardized ratio of weight to height, used as a general indicator of health.
  The Body Mass Index (BMI) is a widely used health indicator. It can be roughly calculated by dividing your body weight (in kilograms) by your height (in meters) squared. If the resulting figure is less than 18.5, you are underweight. A number between 18.5 and 25 indicates a healthy weight. A number above 25 is overweight and a number above 30 is obese. Although the BMI is a generally accepted indicator of health, it is not the only one. For example, a person with a lot of muscle mass can have a high BMI without being in poor health.
Daily calorie intake (DCI) | ONLY ONCE. 10 MINUTES
  An estimate of how many calories the patient must consume in the next 24 hours to maintain their current weight.
  While Basal Metabolic Rate (BMR) is about the number of calories your body needs daily to function effectively when you are at rest, DCI also includes the number of calories you need to function effectively during your daily activities. Thus, to calculate the daily energy needs, two aspects are taken into account:
  Basal Metabolic Rate (BMR): The energy your body needs to maintain basic bodily functions like breathing, heart rate, and temperature regulation, and your Energy for Activity: The energy your body needs to move, depending on your level of physical activity.
Resting heart rate | ONLY ONCE. 10 MINUTES
  Resting heart rate can predict cardiovascular morbidity and mortality. Monitoring heart rate can help in cardiovascular disease prevention and management. The rates of death attributable to cardiovascular disease have declined over the years, yet the burden of disease remains.
  Cardiovascular autonomic neuropathy associated with diabetes mellitus is caused by an impairment of the autonomic system. The prevalence of this condition ranges from 20% to 65%, depending on the duration of the diabetes mellitus. Clinically, the autonomic function disorder is associated with resting tachycardia, exercise intolerance, orthostatic hypotension, intraoperative cardiovascular instability, silent myocardial ischemia and increased mortality.

IPD SHARING:
Plan to Share IPD: Undecided
At the moment the team is working internally to decide what information to share

REFERENCES:
- [Background] Sayer AA, Syddall HE, Dennison EM, Gilbody HJ, Duggleby SL, Cooper C, Barker DJ, Phillips DI. Birth weight, weight at 1 y of age, and body composition in older men: findings from the Hertfordshire Cohort Study. Am J Clin Nutr. 2004 Jul;80(1):199-203. doi: 10.1093/ajcn/80.1.199. PMID 15213049
- [Background] Kim YK, Lee HS, Ryu JJ, In Lee H, Seo SG. Sarcopenia increases the risk for mortality in patients who undergo amputation for diabetic foot. J Foot Ankle Res. 2018 Jun 19;11:32. doi: 10.1186/s13047-018-0274-1. eCollection 2018. PMID 29946364
- [Background] Jimenez S, Rubio JA, Alvarez J, Ruiz-Grande F, Medina C. Trends in the incidence of lower limb amputation after implementation of a Multidisciplinary Diabetic Foot Unit. Endocrinol Diabetes Nutr. 2017 Apr;64(4):188-197. doi: 10.1016/j.endinu.2017.02.009. Epub 2017 Mar 30. English, Spanish. PMID 28417873
- [Result] Li Y, Guo C, Cao Y. Secular incidence trends and effect of population aging on mortality due to type 1 and type 2 diabetes mellitus in China from 1990 to 2019: findings from the Global Burden of Disease Study 2019. BMJ Open Diabetes Res Care. 2021 Nov;9(2):e002529. doi: 10.1136/bmjdrc-2021-002529. PMID 34732399
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Result] Buckinx F, Landi F, Cesari M, Fielding RA, Visser M, Engelke K, Maggi S, Dennison E, Al-Daghri NM, Allepaerts S, Bauer J, Bautmans I, Brandi ML, Bruyere O, Cederholm T, Cerreta F, Cherubini A, Cooper C, Cruz-Jentoft A, McCloskey E, Dawson-Hughes B, Kaufman JM, Laslop A, Petermans J, Reginster JY, Rizzoli R, Robinson S, Rolland Y, Rueda R, Vellas B, Kanis JA. Pitfalls in the measurement of muscle mass: a need for a reference standard. J Cachexia Sarcopenia Muscle. 2018 Apr;9(2):269-278. doi: 10.1002/jcsm.12268. Epub 2018 Jan 19. PMID 29349935
- [Result] Trevino-Aguirre E, Lopez-Teros T, Gutierrez-Robledo L, Vandewoude M, Perez-Zepeda M. Availability and use of dual energy X-ray absorptiometry (DXA) and bio-impedance analysis (BIA) for the evaluation of sarcopenia by Belgian and Latin American geriatricians. J Cachexia Sarcopenia Muscle. 2014 Mar;5(1):79-81. doi: 10.1007/s13539-013-0126-6. Epub 2014 Jan 18. No abstract available. PMID 24442632
- [Result] Han A, Bokshan SL, Marcaccio SE, DePasse JM, Daniels AH. Diagnostic Criteria and Clinical Outcomes in Sarcopenia Research: A Literature Review. J Clin Med. 2018 Apr 8;7(4):70. doi: 10.3390/jcm7040070. PMID 29642478
- [Result] Prior SJ, Ryan AS, Blumenthal JB, Watson JM, Katzel LI, Goldberg AP. Sarcopenia Is Associated With Lower Skeletal Muscle Capillarization and Exercise Capacity in Older Adults. J Gerontol A Biol Sci Med Sci. 2016 Aug;71(8):1096-101. doi: 10.1093/gerona/glw017. Epub 2016 Feb 17. PMID 26888434